CLINICAL TRIAL: NCT04982016
Title: Effects of Preoperative Fluid Therapy on Microcirculatory Reactivity in Patients With MIDCAB After General Anesthesia
Brief Title: Effects of Fluid Therapy on Microcirculatory Reactivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Boqun Cui, Deputy chief physician, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020093X
Record Dates: First submitted 2021-06-24; First posted 2021-07-29 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Microcirculation; Fluid Therapy
Keywords: minimally invasive coronary artery bypass grafting; fuid therapy; microcirculation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): There is no treatment before anesthesia induction.
- Crystal group (Experimental): The fluid reactivity was determined by PLR test before anesthesia induction. The basic value was measured when maintain the head height at 45° for 2 min. and the liquid reactivity value was measured when both legs were raised 45° for 2 min. If △SV >16%, restore the head height to 45°, and 250ml carbonated Ringer's solution was infused (infusion time >10min).
  Interventions: Other: crystal therapy
- Colloidal group (Experimental): The fluid reactivity was determined by PLR test before anesthesia induction. The basic value was measured when maintain the head height at 45° for 2 min. and the liquid reactivity value was measured when both legs were raised 45° for 2 min. If △SV >16%, restore the head height to 45°, and 250ml colloidal fluid was infused (infusion time >10min).
  Interventions: Other: colloid therapy

INTERVENTIONS:
Other: crystal therapy — Infusion of 250ml crystal solution before anesthesia induction
  Arms: Crystal group
Other: colloid therapy — Infusion of 250ml colloid solution before anesthesia induction
  Arms: Colloidal group

SUMMARY:
Through preoperative fluid therapy, to investigate whether it can alleviate the microcirculation dysfunction after induction of anesthesia, and reduce the incidence of perioperative fluid therapy-related complications, thereby accelerating rehabilitation.

DETAILED DESCRIPTION:
Patients undergoing minimally invasive coronary artery bypass graft surgery were randomly divided into crystal group, colloid group and control group. The preoperative fluid reactivity was evaluated according to the passive leg lifting test (PLR). When stroke volume increased (△SV)>16%, the patients in the crystal (carbonate Ringer solution) and the colloid group (hydroxyethyl starch solution) were treated with volume therapy, while the control group was not treated with PLR test and volume therapy. Vascular occlusion test was used to observe the effect of anesthesia induction on tissue oxygen saturation recovery slope (RecStO2) after volume therapy, Goal-directed fluid therapy was used during operation, and the postoperative microcirculation function and the incidence of related complications were observed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Plan to undergo elective minimally invasive coronary artery bypass grafting (left anterior descending branch);
* Sign informed consent

Exclusion Criteria:

* Left ventricular ejection fraction <40%
* Diabetes
* Renal insufficiency (serum creatinine>177umol/L)
* Liver insufficiency (AST, ALT>3 times)
* Peripheral vascular disease
* Carotid artery stenosis (>60%) VOT test contraindications (arm deformity, burns, arteriovenous shunt)
* Use glucocorticoids, vasoactive drugs, inotropic drugs or intra-aortic balloon counterpulsation (IABP)
* Allergic to colloidal fluids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in DesStO2 is assessed | The microcirculation function is measured at 4 time points: patients entered the operating room; 5 minutes after volume therapy; 30 minutes after anesthesia induction; and at the end of the operation
  DesStO2(%/min):The downhill slope of StO2 reflects the oxygen consumption rate
Change in tM is assessed | The microcirculation function is measured at 4 time points: patients entered the operating room; 5 minutes after volume therapy; 30 minutes after anesthesia induction; and at the end of the operation
  The time for minimum value of StO2 to recover to maximum value of StO2

SECONDARY OUTCOMES:
Change in mean arterial pressure is assessed | 4 time points: patients entered the operating room; 5 minutes after volume therapy; 30 minutes after anesthesia induction; and at the end of the operation
Change in heart rate is assessed | 4 time points: patients entered the operating room; 5 minutes after volume therapy; 30 minutes after anesthesia induction; and at the end of the operation
Length of hospital stay | up to 60 days
Duration of stay in the intensive care unit | up to 60 days
Change in HS is assessed | 4 time points: patients entered the operating room; 5 minutes after volume therapy; 30 minutes after anesthesia induction; and at the end of the operation
  HS(ng/ml): As a valuable clinical biomarker for glycocalyx degradation
Change in SDC-1 is assessed | 4 time points: patients entered the operating room; 5 minutes after volume therapy; 30 minutes after anesthesia induction; and at the end of the operation
  SDC-1(ng/ml): As a valuable clinical biomarker for glycocalyx degradation

CONTACTS AND LOCATIONS:
Overall Officials: Boqun Cui, Doctor, Principal Investigator — Anzhen hospital Beijing China